CLINICAL TRIAL: NCT04559191
Title: The Efficacy of Glycemic Control With Continuous Glucose Monitoring on Atheroma Progression: Rationale and Design of the Observation of Coronary Atheroma Progression Under Continuous Glucose Monitoring Guidance in Patients With Type 2 Diabetes Mellitus
Brief Title: Atheroma Progression and Vulnerability Under Continuous Glucose Monitoring
Acronym: OPTIMAL
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cerebral and Cardiovascular Center, Japan (Other)
Responsible Party: Principal Investigator, Yu Kataoka, Chief consultant, National Cerebral and Cardiovascular Center, Japan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M30-152-2
Record Dates: First submitted 2020-09-02; First posted 2020-09-22 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Coronary Atherosclerosis
Keywords: type 2 diabetes mellitus; coronary atherosclerosis; intravascular ultrasound; near-infrared spectroscopy; continuous glucose monitoring
MeSH Terms: conditions — Coronary Artery Disease; Diabetes Mellitus, Type 2 | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- HbA1c-guided group (No Intervention): Glycemic control is controlled by guideline-recommended HbA1c control.
- CGM-guided group (Active Comparator): Glycemic control is controlled by CGM-guided control.
  Interventions: Device: continuous glucose monitoring (CGM)

INTERVENTIONS:
Device: continuous glucose monitoring (CGM) — CGM (FreeStyle Libre Pro®, Abbott, Chicago, Illinoi, the United States)
  Arms: CGM-guided group

SUMMARY:
The OPTIMAL is a single-center, randomized trial to evaluate the efficacy of CGM-based glycemic control on atheroma progression in T2DM patients with CAD by using serial intravascular ultrasound (IVUS) and near-infrared spectroscopy (NIRS) imaging. A total of 90 eligible subjects will be randomized 1:1 into 2 groups to receive either CGM-based glycemic control or HbA1c-baded glycemic management. Coronary angiography and NIRS/IVUS imaging is repeated at the end of the assigned treatment period.

Results: The primary endpoint is the normalized absolute change in total atheroma volume from baseline to 12 months. The secondary endpoints include (1) the absolute change in percent atheroma volume, (2) the percent change in lipid core burden index, (3) the change in coefficient variance measured by CGM, (4) the change in atherogenic markers (high-density lipoprotein functionality, proprotein convertase subxilisin/kexin type 9 and fatty-acid binding proteins), and (5) the frequency of hypoglycemia. Safety will also be evaluated.

DETAILED DESCRIPTION:
Enrollment of 90 patients is planned at National Cerebral & Cardiovascular Center in Japan. Study participants are randomly assigned to either CGM-based glucose management or HbA1c-based glucose management.

Eligible subjects should have CAD requiring elective PCI. HbA1c at screening should be between 7.0 and 10.0%.

Non-culprit vessel with its severe tortuousty and/or calcification will be excluded. Subjects with baseline estimated glomerular filtration rate <40 mL/min/1.73m2 will not be eligible.

After informed consent has been obtained, elective PCI will be conducted to treat culprit lesion. NIRS/IVUS imaging will be conducted to evaluate coronary atheroma.

In the CGM-based glucose management group, CGM (FreeStyle Libre Pro®, Abbott, Chicago, Illinoi, the United States) and HbA1c measurement will be undertaken at baseline and 3, 6, 9 and 12 months following PCI. In the HbA1c-based glucose management group, HbA1c will be measured at baseline and 3, 6, 9 and 12 months after PCI, and CGM will be used at baseline and 12 months in a similar fashion..

With regard to the use of anti-diabetic drugs, in the CGM-guided glycemic control group, endocrinologist will select glucose lowering drugs to fulfill the following CGM-derived goals: (a) the frequency of hypoglycemia=0%, (b) the coefficient of variation <36% and (c) averaged glucose level between 70-180 mg/dl.6 If the frequency of hypoglycemia is over 10% and/or the averaged glucose level is more than 400 mg/dl, patients will be asked to visit within 1 month after CGM measurement. In the HbA1c-guided therapy group, the selection of glucose lowering agents will be made according to the discretion of each endocrinologist to achieve HbA1c <7.0%.

At 12 months following PCI, patients will be hospitalized to take follow-up coronary angiography and intravascular imaging study. NIRS/IVUS imaging in the non-culprit vessel will be conducted again in a similar fashion.

ELIGIBILITY:
Inclusion Criteria:

* Male of female between 20 and 85 years of age
* Type 2 diabetic patients with coronary artery disease who require PCI
* The presence of mild stenosis in the non-target vessel (% diameter stenosis between 10-50%)
* 7.0 ≤ HbA1c ≤ 10.0%
* HbA1c ≤ 10.0% in subjects who receive insulin, sulfonylurea or nateglinide
* Ability to understand the requirements of the study and to provide informed consent

Exclusion Criteria:

* very tortuous coronary artery and/or severe calcification which is unsuitable for intravascular imaging
* Subjects with severe renal dysfunction (estimated glomerular filtration rate < 40 mL/min/1.73m2)
* the absence of any atherosclerotic lesions in the non-target vessel those who take PCSK9 inhibitor
* current enrolment in another investing device or drug study pregnancy

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
the normalized absolute change in total atheroma volume on serial intravascular ultrasound imaging. | from baseline to 12 months
  This measure is analyzed by serial intravascular ultrasound imaging.

SECONDARY OUTCOMES:
the absolute change in percent atheroma volume on serial intravascular ultrasound imaging. | from baseline to 12 months
  This measure is analyzed by serial intravascular ultrasound imaging.
the percent change in lipid core burden index on serial near-infrared spectroscopy imaging. | from baseline to 12 months
  This measure is analyzed by serial near-infrared spectroscopy imaging.
the change in coefficient variance evaluated by CGM | from baseline to 12 months
  This measure is analyzed by CGM.
the correlation of change in concentration of serum proprotein convertase subxilisin/kexin type 9 with the normalized absolute change in total atheroma volume | from baseline to 12 months
  The correlation of IVUS measure with concentration of serum proprotein convertase subxilisin/kexin type 9 is analyzed.
change in TAV under the use of specific anti-diabetic agents (dipeptidyl peptidase-4 inhibitors, sodium-glucose transport protein 2 inhibitors and glucagon-like peptide-1 agonists) | from baseline to 12 months
  This measure is analyzed by serial intravascular ultrasound imaging.
the frequency of hypoglycemia | from baseline to 12 months
  This event is collected through each clinical visit.

CONTACTS AND LOCATIONS:
Overall Officials: Yu Kataoka, MD, Principal Investigator — National Cerebral & Cardiovascular Center
Locations (1):
- National Cerebral & Cardiovascular Center, Suita, Japan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Kataoka Y, Hosoda K, Makino H, Matsubara M, Matsuo M, Ohata Y, Koezuka R, Tamanaha T, Tomita T, Honda-Kohmo K, Noguchi M, Son C, Nishimura K, Asaumi Y, Miyamoto Y, Noguchi T, Yasuda S. The efficacy of glycemic control with continuous glucose monitoring on atheroma progression: rationale and design of the Observation of Coronary Atheroma Progression under Continuous Glucose Monitoring Guidance in Patients with Type 2 Diabetes Mellitus (OPTIMAL). Cardiovasc Diagn Ther. 2019 Oct;9(5):431-438. doi: 10.21037/cdt.2019.09.02. PMID 31737515